CLINICAL TRIAL: NCT06503718
Title: Management of Closed Diaphyseal Displaced Leg Fractures in Children and Adolescents: Should Osteosynthesis Be Favored From the Start?
Brief Title: Management of Closed Diaphyseal Displaced Leg Fractures in Children and Adolescents
Acronym: FFD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9244
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Tibial Fractures
Keywords: Tibial Fractures; Osteosynthesis, Fracture; Closed Fracture
MeSH Terms: conditions — Tibial Fractures; Fractures, Bone; Fractures, Closed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most displaced tibial shaft fractures in pediatric patients have traditionally been treated after reduction by cast immobilization with good long-term results. Recently, there has been a growing trend towards surgical intervention by osteosynthesis from the outset. This study aims to describe the results of orthopedic treatment and osteosynthesis from the outset.

ELIGIBILITY:
Inclusion Criteria:

* Minor subject (under 18 years old)
* Subject treated at the HUS, between June 1, 2004 and April 31, 2024, for a fracture of the displaced diaphysis of the tibia treated orthopedically or by osteosynthesis reviewed after more than 6 months
* Absence of written opposition in the medical file of the subject (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.

Exclusion criteria:

* Presence of opposition from the subject (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.
* Non-displaced and/or displaced fracture not located at the level of the tibial diaphysis
* Open fracture
* Incomplete or unusable file

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor subject (under 18 years old) treated at the HUS, between June 1, 2004 and April 31, 2024, for a fracture of the displaced diaphysis of the tibia treated orthopedically or by osteosynthesis reviewed after more than 6 months
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the result of orthopedic treatment and osteosynthesis from the outset | Up to 6 months
  Use of the functional score for this assessment :
  Scores :
  * 95-100 : Excellent
  * 75-94 : Good
  * 51-74 : Fair
  * 0-50 : Poor

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Pédiatrique - CHU de Strasbourg - France, Strasbourg, France